CLINICAL TRIAL: NCT06579521
Title: Connecting Alcohol Myopia to Real-World Risk Behaviors Through Cognitive Ecological Momentary Assessment (REACT Phase II: Lab and EMA)
Brief Title: Real-world Experiences of Alcohol and Cognitions Over Time
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anna Jaffe, Associate Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00018677; R21AA029489 (NIH)
Record Dates: First submitted 2024-08-15; First posted 2024-08-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alcohol (Experimental)
  Interventions: Other: Alcohol

INTERVENTIONS:
Other: Alcohol — A standard dose of alcohol will be administered (volume calculated with regard to age, sex assigned at birth, height, and weight) in the form of vodka and combined with mixer at a 1:4 ratio to reach a target breath alcohol concentration of .08%.

SUMMARY:
The goal of this clinical trial is to examine how alcohol affects young adults' attention in both laboratory and real-world settings through phone-based cognitive tasks. The main questions this trial is designed to answer are:

* How well do the phone-based cognitive tasks capture alcohol's effects on attention?
* Does the effect of alcohol on attention contribute to risk-taking?

Participants will complete cognitive tasks to assess attention before and after consuming a standard amount of alcohol in the laboratory, and during surveys completed through a phone app for eight weekends.

DETAILED DESCRIPTION:
The goal of this study is to develop cognitive tasks that assess alcohol-related attentional narrowing (i.e., alcohol myopia) for smartphone-based ecological momentary assessment (EMA). In Phase I, tasks were adapted from computer to smartphone format and refined through interviews with young adults who provided feedback on mock-ups. In Phase II (the current trial), feasibility, acceptability, reliability, and validity of the adapted tasks will be tested in lab and EMA. Young adults who pass an online pre-screening and phone screening will complete an initial lab session involving self-report questionnaires, alcohol consumption (target breath alcohol concentration [BrAC] = .08%), and general cognitive and myopia-specific tasks. All participants in Phase II will be assigned to receive a dose of alcohol in the lab session; task performance will be compared within individuals from before to after they are intoxicated. Participants will remain in the lab until their BrAC reduces to a level of .03% and they can pass a field sobriety test. These same participants will then complete EMA while wearing transdermal alcohol biosensors for 8 consecutive weekends, including one morning survey and at least two evening surveys per day. Then, participants will return to the lab for a follow-up session involving self-report questions and an interview eliciting additional feedback. Findings will help to clarify the role of alcohol myopia as a mechanism linking intoxication to real-world risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* aged 21-25
* drink at least 2x/week in the past month
* at least 1 past-month heavy episodic drinking event (4+/5+ standard drinks in a day for females/males)
* have an iPhone
* able to read and understand English
* willing to complete all study procedures

Exclusion Criteria:

* history of alcohol-related treatment or hospitalization
* medical contraindications for alcohol consumption (e.g., contraindicated medication, major psychiatric illness, history of seizure, gastric bypass surgery, cardiac pacemaker, major illness such as liver cirrhosis or hepatitis, past traumatic brain injury, asthma exacerbated by alcohol use, consistent flushing response to alcohol use) or pregnancy, nursing an infant, or plans to become pregnant in the next 8 weeks (i.e., during the EMA monitoring period)
* substantial visual impairment or color blindness (given that cognitive tasks rely on visual cues)

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-08-18 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Central Counting Task (phone) | Baseline and after alcohol consumption in the laboratory (an average of approximately 1 hour after baseline)
  On a phone, participants will count the number of times a crosshair flashes in the center of the screen. Each trial will include between 1 and 4 flashes. There will be 6 trials per block. After a training block, there will be two blocks administered while sober. After alcohol consumption, three blocks will be administered on the ascending limb of the BrAC curve. Number of accurate responses will be evaluated.
Peripheral Probe Identification Task (phone) | Baseline and after alcohol consumption in the laboratory (an average of approximately 1 hour after baseline)
  While counting the number of times a crosshair flashes in the center of a phone screen (central counting task), participants will also be asked to monitor a cued corner (if possible), and shown an array of four colored stimuli. In each trial, they will be asked to identify whether the color of a probe matches the cued stimulus, with a 50% likelihood of matching. After a training block, there will be two blocks administered while sober. After alcohol consumption, three blocks will be administered on the ascending limb of the BrAC curve. Number of accurate responses will be evaluated.
Visual Categorization Task (phone) | Baseline and after alcohol consumption in the laboratory (an average of approximately 1 hour after baseline)
  On a phone, participants will be presented with one of two visual stimuli (shapes) in a random sequence with equal probability, and asked to categorize each stimuli as quickly as possible (e.g., "Is this a square or circle?") with placement of response buttons (right or left side of screen) randomized. Each trial consists of a shape categorization. There are 12 trials per block. After a training block, there will be two blocks administered while sober. After alcohol consumption, three blocks will be administered on the ascending limb of the BrAC curve. Differences in response time will be evaluated for one-back stimuli (change vs. no change) and two-back stimuli (change vs. no change).

SECONDARY OUTCOMES:
Central Counting Task (desktop) | Baseline and after alcohol consumption in the laboratory (an average of approximately 1 hour after baseline)
  On a phone, participants will count the number of times a crosshair flashes in the center of the screen. Each trial will include between 1 and 4 flashes. A training block of 12 trials will be administered while sober. After alcohol consumption, two blocks of 120 trials each will be administered on the ascending limb of the BrAC curve. Number of accurate responses will be evaluated.
Peripheral Probe Identification Task (desktop) | Baseline and after alcohol consumption in the laboratory (an average of approximately 1 hour after baseline)
  While counting the number of times a crosshair flashes in the center of a desktop screen (central counting task), participants will also be asked to monitor a cued corner (if possible), and shown an array of four colored stimuli. In each trial, they will be asked to identify whether the color of a probe matches the cued stimulus, with a 50% likelihood of matching. A training block of 12 trials will be administered while sober. After alcohol consumption, two blocks of 120 trials each will be administered on the ascending limb of the BrAC curve. Number of accurate responses will be evaluated.
Auditory Categorization Task (desktop) | Baseline and after alcohol consumption in the laboratory (an average of approximately 1 hour after baseline)
  On a desktop, participants will be presented with one of two auditory stimuli (high and low tones) in a random sequence with equal probability, and asked to categorize each stimuli as quickly as possible with placement of response options (shown on right or left side of screen) randomized. Each trial consists of a shape categorization. A training block of 12 trials will be administered while sober. After alcohol consumption, five blocks of 100 trials each will be administered on the ascending limb of the BrAC curve. Differences in response time will be evaluated for one-back stimuli (change vs. no change) and two-back stimuli (change vs. no change).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share limited, de-identified datasets for the purposes of data analysis and dissemination.
Time Frame: During data collection, data will be submitted biannually to the NIMH Data Archive.
Access Criteria: Individual requests to access data with intended purpose should be made to Dr. Jaffe and will be reviewed by the investigative team. Requests can also be made through the NIMH Data Archive